CLINICAL TRIAL: NCT07005570
Title: Short-Course Radiotherapy Followed by Sequential Chemotherapy Combined With PD-1 Monoclonal Antibody and Bevacizumab Versus Short-Course Radiotherapy Followed by Sequential Chemotherapy as Total Neoadjuvant Therapy in pMMR/MSS Locally Advanced Rectal Cancer
Brief Title: Short-course Radiotherapy Followed by Sequential Chemotherapy With or Without PD-1 Monoclonal Antibody and Bevacizumab as Total Neoadjuvant Therapy in pMMR/MSS Locally Advanced Rectal Cancer （SPARK）
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dechang Diao (Other)
Responsible Party: Sponsor-Investigator, Dechang Diao, PH.D., Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-288
Record Dates: First submitted 2025-05-10; First posted 2025-06-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: pMMR/MSS Locally Advanced Rectal Cancer
Keywords: PD-1 monoclonal antibody; VEGF monoclonal antibody; total neoadjuvant therapy (TNT); pMMR/MSS locally advanced rectal cancer
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Short-course radiotherapy → CAPOX regimen chemotherapy (6 cycles) → undergo surgery or watch-and-wait strategy within 2-4 weeks after the last dose of capecitabine.
  Interventions: Other: Short-course radiotherapy followed by sequential chemotherapy
- Experimental group (Experimental): Short-course radiotherapy → PD-1 monoclonal antibody and bevacizumab combined with CAPOX regimen chemotherapy (4 cycles) → PD-1 monoclonal antibody combined with CAPOX regimen chemotherapy (2 cycles) → undergo surgery or watch-and-wait strategy within 2-4 weeks after the last dose of capecitabine.
  Interventions: Other: Short-course radiotherapy followed by sequential chemotherapy combined with PD-1 monoclonal antibody and bevacizumab

INTERVENTIONS:
Other: Short-course radiotherapy followed by sequential chemotherapy combined with PD-1 monoclonal antibody and bevacizumab — Short-course radiotherapy → PD-1 monoclonal antibody and bevacizumab combined with CAPOX regimen chemotherapy (4 cycles) → PD-1 monoclonal antibody combined with CAPOX regimen chemotherapy (2 cycles) → undergo surgery or watch-and-wait strategy within 2-4 weeks after the last dose of capecitabine.
  Arms: Experimental group
Other: Short-course radiotherapy followed by sequential chemotherapy — Short-course radiotherapy → CAPOX regimen chemotherapy (6 cycles) → undergo surgery or watch-and-wait strategy within 2-4 weeks after the last dose of capecitabine.
  Arms: Control group

SUMMARY:
Safety and efficacy of Short-Course Radiotherapy Followed by Sequential Chemotherapy with or without PD-1 Monoclonal Antibody and Bevacizumab as Total Neoadjuvant Therapy in pMMR/MSS Locally Advanced Rectal Cancer.

Complete Response (CR) Rate of Short-Course Radiotherapy Followed by Sequential Chemotherapy with or without PD-1 Monoclonal Antibody and Bevacizumab as Total Neoadjuvant Therapy in pMMR/MSS Locally Advanced Rectal Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed written informed consent form.
2. Age ≥18 and ≤75 years at enrollment.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
4. Life expectancy >2 years.
5. Histologically confirmed rectal adenocarcinoma.
6. Tumor biopsy demonstrating pMMR (all four mismatch repair proteins-MSH1, MSH2, MSH6, and PMS2-positive by immunohistochemistry) or genetic testing confirming MSS (microsatellite stable).
7. Clinical stage II-III rectal cancer (cT3-4NanyM0 or cTxN+M0) per AJCC 8th Edition TNM staging, assessed via high-resolution MRI ± endoscopic ultrasound/transrectal Doppler ultrasound. Tumor must be ≤12 cm from the anal verge by MRI.
8. Pre-enrollment surgical evaluation by an attending surgeon confirming eligibility for curative-intent R0 resection.
9. No prior systemic or local anti-cancer therapy for rectal cancer (radiotherapy, chemotherapy, immunotherapy, biologics, or small-molecule targeted therapy).
10. Willingness to provide tumor tissue (archival or fresh biopsy) and peripheral blood samples for biomarker analysis during screening and study procedures.
11. Adequate organ function.
12. For women of childbearing potential (WOCBP):Negative urine or serum pregnancy test within 3 days prior to treatment (serum test required if urine result is inconclusive).Agreement to use highly effective contraception (e.g., intrauterine device, hormonal implants) from screening until 120 days after last study treatment. Periodic abstinence and calendar-based methods are prohibited.
13. The subject is willing and able to comply with scheduled visits, treatment regimens, laboratory tests, and other study requirements as outlined in the protocol.

Exclusion Criteria:

1. Suspected metastatic lesions or locally advanced unresectable disease regardless of stage.
2. History of other malignancies within 5 years prior to enrollment, except those cured by local therapy (e.g., basal/squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the breast).
3. Concurrent participation in another interventional clinical trial (observational or non-interventional studies allowed).
4. Acute complications requiring emergency surgery (e.g., bowel obstruction, perforation, hemorrhage).
5. Multiple primary rectal cancers.
6. Prior pelvic/abdominal radiotherapy.
7. Conditions impairing oral drug absorption (e.g., dysphagia, malabsorption syndrome).
8. Prior systemic/local anti-tumor therapy for locally advanced rectal cancer (surgery, chemotherapy, radiotherapy, immunotherapy [checkpoint inhibitors/agonists, cell therapy], biologics, or targeted agents).
9. Non-specific immunomodulators (e.g., interleukins, interferons) within 2 weeks or anti-tumor herbal medicines within 1 week prior to treatment.
10. Active autoimmune disease requiring systemic immunosuppression (e.g., corticosteroids >10 mg/day prednisone equivalent) within 2 years (hormone replacement allowed).
11. History of non-infectious pneumonitis or interstitial lung disease requiring steroids.
12. Bleeding diathesis/coagulopathy or chronic anticoagulation (e.g., CHADS2 score ≥2 for atrial fibrillation).
13. Uncontrolled comorbidities (e.g., decompensated cirrhosis, nephrotic syndrome, peptic ulcers) or psychiatric disorders affecting consent/study compliance.
14. Cardiac history:Myocarditis/cardiomyopathy/malignant arrhythmias.Unstable angina/CHF within 12 months.Arterial thromboembolism within 6 months (e.g., stroke, TIA).Grade ≥3 venous thromboembolism (CTCAE v5.0).Uncontrolled hypertension (SBP ≥160 mmHg/DBP ≥100 mmHg).
15. Active inflammatory bowel disease (Crohn's/ulcerative colitis) or chronic diarrhea.

16Active severe infection requiring hospitalization/systemic antibiotics within 4 weeks (excluding HBV/HCV antivirals).

17.Major surgery/trauma within 30 days or minor procedures within 3 days (excluding PICC placement).

18.Immunodeficiency (HIV-positive, chronic immunosuppressants). 19.Active tuberculosis (confirmed by sputum/X-ray) or syphilis. 20.Prior allogeneic organ/stem cell transplantation. 21.Active hepatitis:HBV: HBsAg+ with HBV-DNA >1000 copies/mL (200 IU/mL) without antiviral therapy.HCV: Anti-HCV+ with detectable HCV-RNA.

22.Live vaccines within 30 days or planned during study. 23.Hypersensitivity to study drugs/monoclonal antibodies. 24.Substance abuse or psychiatric disorders compromising compliance. 25.Pregnancy/lactation. 26.Conditions confounding efficacy/safety assessments or limiting survival evaluation (e.g., leukemoid reaction [WBC >20×10⁹/L], cachexia [>10% weight loss in 3 months], BMI ≤18).

27.Other conditions deemed inappropriate by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate | 2-4week
  Defined as the proportion of subjects achieving pathological complete response (pCR) or clinical complete response (cCR) following neoadjuvant therapy. pCR is characterized by the absence of residual tumor in the resected primary tumor site and lymph nodes; cCR is defined as achieving ycT0N0 status according to the 2024 CWWD criteria.
Adverse events | 2-4week
  Incidence and severity of adverse events according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Dechang Diao, Dr, Study Director — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No